CLINICAL TRIAL: NCT03201497
Title: Prospective Registration of Severe Pneumocystis Jiroveci Pneumonia Requiring ICU
Brief Title: Prospective Registration of Severe Pneumocystis Jiroveci Pneumonia Requiring ICU Admission
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PJP2017-1
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Pneumocystis Jiroveci Pneumonia; Intensive Care Unit
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with PJP: PJP patients in ICU with or without HIV infection

SUMMARY:
the investigators aim to set up a multicenter registry study for severe PJP requiring ICU admission. The purpose of this study is

1. to establish a prospective severe PJP registry about clinical characteristics, laboratory and radiographic findings, critical care management and outcomes.
2. to explore the predictive factors associated with outcomes ;
3. to compare the difference between PJP patients with HIV and without HIV infection.

DETAILED DESCRIPTION:
Pneumocystis jiroveci pneumonia (PJP) is a common opportunistic infection in immunocompromised patients. Although the mortality of patients with mild to moderate PJP has declined substantially, the reported outcomes of severe PJP requiring ICU admission, especially with mechanical ventilation are grave. The data on this group of patients is very limited and mainly comes from retrospective studies.

the investigators aim to set up a multicenter registry study for patient with severe PJP requiring ICU admission to provide comprehensive descriptive data on diagnosis, clinical course, critical care management and outcomes in a large cohort.

All patients with PJP admitted to the participating ICU during a two-year period will be enrolled. The CRF will be made available to the participating sites as a printable paper-based CRF.

The following individual patient data for study participants will be collected:

* General demographic information
* Presence of risk factors for PJP and comorbid condition
* use of prophylactic SMZ/TMP, immunosuppressive medications prior to ICU admission
* Information about PJP and co-infection diagnosis
* vital signs, laboratory(blood serum and BALF sample) and radiologic data at ICU admission and during ICU stay
* organ failures and severity of the disease at admission, new onset of organ failures during ICU stay
* Medications for PJP, time course and modalities and settings for respiratory support
* ICU, 28-day mortality, hospital, 90-day mortality

ELIGIBILITY:
Inclusion Criteria:

* diagnosis with PJP, confirmed by PCR or methenamine silver stain of sample from BALF, aspirate or sputum;
* ICU admission due to PJP-related respiratory failure

Exclusion Criteria:

* NO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PJP patients requiring ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
28-day ICU mortality | Day 28
  28 days mortality after ICU admission

SECONDARY OUTCOMES:
hospital mortality | Day 90 (censored at hospital discharge if discharge prior to Day 90)
  mortality at hospital discharge
ICU length of stay | Day 90
  ICU length of stay at ICU discharge
hospital length of stay | Day 90
  hospital length of stay at hospital discharge
occurrence of SMZ/TMP treatment failure | day 7 after SMZ/TMP treatment
  SMZ/TMP treatment failure is defined as worsening P/F or radiographic features with a requirement for an increased respiratory support after 7 days of SMZ/TMP treatment (SMZ/TMP)
mechanical ventilation free days | day 28
  days without mechanical ventilation during ICU
occurrence of non-invasive mechanical ventilation | day 28
  Non-invasive mechanical ventilation failure is defined as need for switch from non-invasive mechanical ventilation to invasive mechanical ventilation due to deteriorated respiratory failure
occurrence of pneumothorax or pneumomediastinum | day 28
  pneumothorax or pneumomediastinum is confirmed by chest X ray or CT
ICU acquired infectious disease | day 28
  incidence of pulmonary of extra-pulmonary infections. Diagnosis of infections disease will be defined by the need of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, Dr, Study Director — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: Undecided